CLINICAL TRIAL: NCT02344108
Title: A Pilot Study to Evaluate the Safety and Efficacy of the Hypoglossal Nerve Stimulator in Adolescents and Young Adults With Down Syndrome and Obstructive Sleep Apnea
Brief Title: A Pilot Study to Evaluate the Hypoglossal Nerve Stimulator in Adolescents With Down Syndrome and Obstructive Sleep Apnea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Christopher Hartnick, M.D. (Other)
Collaborators: Emory University (Other); Children's Hospital Medical Center, Cincinnati (Other); Inspire Medical Systems, Inc. (Industry); University of Pittsburgh (Other); Children's Hospital of The King's Daughters (Other)
Responsible Party: Sponsor-Investigator, Christopher Hartnick, M.D., Principal Investigator, Massachusetts Eye and Ear Infirmary
Organization: Massachusetts Eye and Ear Infirmary (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14-146H; 2019P001786 (Other: Partners Human Research Committee)
Record Dates: First submitted 2015-01-13; First posted 2015-01-22 (Estimated); Results first posted 2022-02-11 (Actual); Last update posted 2022-04-12 (Actual); Status verified 2022-04

CONDITIONS: Sleep Apnea, Obstructive; Down Syndrome
MeSH Terms: conditions — Sleep Apnea, Obstructive; Down Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Inspire® Upper Airway Simulation System (Experimental): Subjects meeting inclusion criteria, including sleep study and drug induced sleep endoscopy criteria, will undergo surgical placement of a hypoglossal nerve simulator (Inspire® Upper Airway Simulation System Model 3028 IPG). The simulator will be activated one month after surgery and subjects will undergo repeat sleep study evaluation and device titration at one, two, six and twelve months after implantation. Subjects will be followed for one year to determine safety and efficacy of the device.
  Interventions: Device: Inspire® Upper Airway Simulation System (Model 3028 IPG )

INTERVENTIONS:
Device: Inspire® Upper Airway Simulation System (Model 3028 IPG ) — Subjects will be implanted with a hypoglossal nerve stimulator. Safety and efficacy of implantation will be evaluated.
  Other Names: hypoglossal nerve stimulator

SUMMARY:
Obstructive sleep apnea (OSA) affects up to 1% of the general pediatric population and is associated with adverse behavior and quality of life, as well as long term cardiopulmonary system complications. Trisomy 21 (Down Syndrome) is the most common chromosomal disorder, with a incidence of approximately 1 per 660-800 births. Patients with Down Syndrome have a higher incidence of OSA than the general pediatric population, with rates of 30-60%, resulting in increased morbidity and decreased quality of life for affected individuals. In children, adenotonsillectomy (T&A) is often a contributing factor to OSA, and adenotonsillectomy is a first line treatment. Children with Down Syndrome often undergo T&A for obstructive sleep apnea, however 30-50% will have persistent obstructive sleep patterns requiring continuous positive pressure airway support (CPAP) or tracheotomy. Persistent obstruction is attributed to anatomic and physiologic differences in this population, including reduced muscular tone, macroglossia, maxillary hypoplasia, and lingual tonsil hypertrophy. This pilot study is designed to determine if the Inspire® Upper Airway Simulation System, Model 3024 IPG, and any subsequent iteration thereof that are approved under P130008 for the treatment of obstructive sleep apnea, which has already been approved for use in adults with OSA, can be safely implanted and used in adolescents and young adults with Down Syndrome.

DETAILED DESCRIPTION:
The study will be a multi-center, prospective, single-arm study conducted under a common implant and follow-up protocol. Twenty-one adolescents and young adults (10-21 years of age) with Down Syndrome with moderate to severe obstructive sleep apnea after adenotonsillectomy will be identified through a Multi-Disciplinary clinic for patients with Trisomy 21 at each of our participating sites Patients and their parents will be screened by a senior pulmonologist and pediatrician for medical clearance and willingness to participate. Subjects will then undergo preoperative evaluation with an in-lab polysomnogram (PSG), evaluation by a pediatric otolaryngology surgeon, and drug induced sleep endoscopy (DISE) to ensure all inclusion and exclusion criteria are met. Subjects meeting eligibility criteria will then be implanted with the Inspire® Upper Airway Simulation System, Model 3024 IPG, and any subsequent iteration thereof that are approved under P130008 for the treatment of obstructive sleep apnea, a hypoglossal nerve stimulator, after informed consent. Surgery will be performed by senior pediatric otolaryngologists who have completed a training program for the Inspire® system. Subjects will then adhere to a follow-up schedule. The device will be activated and settings titrated during an in-lab sleep study 1 month postoperatively. Quality of life surveys and device interrogation will be conducted at timed intervals. Subjects will then undergo in-lab polysomnography at 2 months, 6 months, and 12-months, then on an annual basis, and the device titrated as needed. All personnel adjusting device parameters will be trained in programming the Inspire® system. For this pilot study, we will evaluate safety and efficacy over the first year after device implantation.

ELIGIBILITY:
Inclusion Criteria:

* Only children and young adults with Down Syndrome age 10-21 years with prior adenotonsillectomy will be considered for the study.
* Subjects must have BMI <95th percentile for age
* All subjects must have moderate to severe OSA (AHI >10, AHI <50, no more than 25% AHI attributable to central events) based on prior in-lab polysomnography performed after adenotonsillectomy.
* Subjects must have either tracheotomy or be ineffectively treated with CPAP due to noncompliance, discomfort, un-desirable side effects, persistent symptoms despite compliance use, or refusal to use the device.
* Children and their parents must be willing to have stimulation hardware permanently implanted, and be willing to participate in follow-up visits, postoperative polysomnography, and questionnaire completion.
* Children's parents must complete a questionnaire confirming that their child is capable of communicating feelings of pain or discomfort. They must also confirm they are able to assess their child for adverse effects related to device implantation.
* Children and their parents must be proficient in English for this pilot study in order to ensure full disclosure during the consent process, as well as have the ability to communicate with all staff, at all times, regarding any questions about participation or concerns about this device.
* In order to participate, subjects will require written consent from both parents. All study subjects must provide written assent as well.

Exclusion Criteria:

* Subjects will be excluded if they meet the following criteria: BMI >95th percentile for age, apnea hypopnea index (AHI) <10 or >50 on in-lab polysomnography (PSG), central or mixed apneas accounting for >25% of the total AHI, any anatomic finding on physical exam or drug induced sleep endoscopy (DISE) that would compromise the performance of stimulation (e.g. concentric soft palate collapse), other medical conditions resulting in medical instability (e.g. congestive heart failure, recent open heart surgery, immunosuppression, or chronic lung disease or aspiration), presence of another medical condition requiring future magnetic resonance imaging (MRI), history of cholesteatoma, or patients with another implantable device which could interact unintentionally with the Inspire system.
* Subjects in whom general anesthesia for a surgical procedure is contraindicated due to other medical illnesses or conditions will be excluded.
* Subjects with a life expectancy < 12 months will be excluded.
* Subjects who are unable to communicate pain or discomfort to their caretaker/parent, based on parental or investigator assessment, will be excluded.
* Subjects with a history of bleeding or clotting disorders and those on blood thinning or NSAID medications will be excluded from participation.
* Subjects taking muscle relaxant medication will be excluded from participation.
* Female subjects who are pregnant or plan to become pregnant during the study period will be excluded. All female subjects will undergo urine beta-HCG testing on the day of procedures requiring general anesthesia (DISE, implantation, and any other unanticipated surgical procedures related to implantation). Subjects who are positive will not undergo surgical implantation or procedures under general anesthesia.
* Subjects deemed unfit for participation by investigators or any other reason will be excluded.

Ages: 10 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 42 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2021-07-23 (Actual); Study Completion 2021-09-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher J Hartnick, MD, Principal Investigator — Massachusetts Eye and Ear
Locations (5):
- United States (5):
  - Children's Healthcare of Atlanta - Egleston Hospital, Atlanta, Georgia
  - Massachusetts Eye and Ear, Boston, Massachusetts
  - Cincinnati Children's Hospital, Cincinnati, Ohio
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Children's Hospital of The King's Daughters, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yu PK, Stenerson M, Ishman SL, Shott SR, Raol N, Soose RJ, Tobey A, Baldassari C, Dedhia RC, Pulsifer MB, Grieco JA, Abbeduto LJ, Kinane TB, Keamy DG Jr, Skotko BG, Hartnick CJ. Evaluation of Upper Airway Stimulation for Adolescents With Down Syndrome and Obstructive Sleep Apnea. JAMA Otolaryngol Head Neck Surg. 2022 Jun 1;148(6):522-528. doi: 10.1001/jamaoto.2022.0455. PMID 35446411
- [Derived] Stenerson ME, Yu PK, Kinane TB, Skotko BG, Hartnick CJ. Long-term stability of hypoglossal nerve stimulation for the treatment of obstructive sleep apnea in children with Down syndrome. Int J Pediatr Otorhinolaryngol. 2021 Oct;149:110868. doi: 10.1016/j.ijporl.2021.110868. Epub 2021 Aug 5. PMID 34371294
- [Derived] Jayawardena ADL, Randolph GW, Hartnick CJ. Pediatric Modifications to Hypoglossal Nerve Stimulation for Obstructive Sleep Apnea: How I Do It. Laryngoscope. 2021 Feb;131(2):423-424. doi: 10.1002/lary.28661. Epub 2020 Apr 9. No abstract available. PMID 32271464
- [Derived] Caloway CL, Diercks GR, Keamy D, de Guzman V, Soose R, Raol N, Shott SR, Ishman SL, Hartnick CJ. Update on hypoglossal nerve stimulation in children with down syndrome and obstructive sleep apnea. Laryngoscope. 2020 Apr;130(4):E263-E267. doi: 10.1002/lary.28138. Epub 2019 Jun 20. PMID 31219619
- [Derived] Diercks GR, Wentland C, Keamy D, Kinane TB, Skotko B, de Guzman V, Grealish E, Dobrowski J, Soose R, Hartnick CJ. Hypoglossal Nerve Stimulation in Adolescents With Down Syndrome and Obstructive Sleep Apnea. JAMA Otolaryngol Head Neck Surg. 2018 Jan 1;144(1):37-42. doi: 10.1001/jamaoto.2017.1871. PMID 29098288
- [Derived] Diercks GR, Keamy D, Kinane TB, Skotko B, Schwartz A, Grealish E, Dobrowski J, Soose R, Hartnick CJ. Hypoglossal Nerve Stimulator Implantation in an Adolescent With Down Syndrome and Sleep Apnea. Pediatrics. 2016 May;137(5):e20153663. doi: 10.1542/peds.2015-3663. PMID 27244805

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited by their local otolaryngologist-investigator, many of whom were referred by Down syndrome clinical programs and other providers. National Down syndrome organizations assisted with study advertisements.
Pre-assignment Details: Enrollment in this study was defined at the time the informed consent forms were signed. Following enrollment, patients underwent drug-induced sleep endoscopies (DISEs) and baseline polysomnography (PSG) unless, per protocol, these procedures had been completed within a set time from enrollment. Patient medical records were reviewed in detail, along with the baseline DISE and PSG results, to confirm eligibility prior to scheduling hypoglossal nerve stimulator implantation.
Groups:
- Inspire® Upper Airway Simulation System: Subjects meeting inclusion criteria, including sleep study and drug induced sleep endoscopy criteria, underwent surgical placement of a hypoglossal nerve simulator (Inspire® Upper Airway Simulation System Model 3028 IPG). The simulator was activated one month after surgery and subjects underwent repeat sleep study evaluation and device titration at one, two, six and twelve months after implantation. Subjects were followed for one year to determine safety and efficacy of the device.
Period: Overall Study
Arm/Group | Inspire® Upper Airway Simulation System
Started | 42
Completed | 42
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Only participants who underwent hypoglossal nerve stimulator implantation are included here in the baseline analysis.
Arm/Group | Inspire® Upper Airway Simulation System
Number analyzed (Participants) | 42
Age, Customized [Count of Participants; unit: Participants]
  Age range: 10 to 13 years old | 13
  Age range: 14 to 17 years old | 19
  Age range: 18 to 21 years old | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 38
  Unknown or Not Reported | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 40
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States: Massachusetts Eye and Ear, Boston, MA | 25
  United States: Cincinnati Children's Hospital Medical Center, Cincinnati, OH | 8
  United States: Children's Hospital of Atlanta, Atlanta, GA | 4
  United States: Children's Hospital of Pittsburgh, Pittsburgh, PA | 3
  United States: Eastern Virginia Medical School, Norfolk, VA | 2
Baseline OSA-18 total survey score [Mean (Standard Deviation); unit: units on a scale] — The OSA-18 generates from participant responses a total score between 18 and 126 which is designed to reflect the impact of obstructive sleep apnea on the pediatric patient's quality of life. Higher total scores on the OSA-18 indicate a greater, negative impact on quality of life; while lower scores indicate a lesser impact on quality of life. Interpretation of total scores is as follows: minimal OSA impact for scores under 60; moderate OSA impact for scores between 60 and 80; and severe OSA impact for scores above 80.
  units on a scale | 66.0 (19.8)
Baseline OSA-18 overall quality of life score [Mean (Standard Deviation); unit: units on a scale] — The OSA-18 questionnaire includes a stand-alone question that asks to rate the child's overall quality of life on a scale from 0 (indicating worst quality of life possible) to 10 (indicating best quality of life possible).
  units on a scale | 5.1 (2.0)
Baseline Epworth Sleepiness Scale (ESS) survey score [Mean (Standard Deviation); unit: units on a scale] — The ESS is a validated survey of daytime sleepiness. The ESS is scored as the sum of all items with scores ranging from 0 to 24 and higher scores indicating worse symptoms.
  units on a scale | 10.0 (7.3)
Baseline apnea-hypopnea index (AHI) [Mean (Standard Deviation); unit: events per hour] — The apnea-hypopnea index (AHI) is a measure of the number of times per hour that an apnea or hypopnea event occurs during sleep. Apneas are defined as short pauses in breathing, while hypopnea is defined as shallow breathing. The AHI is useful in evaluating obstructive sleep apnea (OSA). The normal pediatric range is typically defined as an AHI of less than 1 event per hour. An AHI between 5 and 10 events per hour is consistent with moderate OSA, while an AHI above 10 suggests severe OSA.
  events per hour | 23.5 (9.7)
Baseline obstructive apnea-hypopnea index [Mean (Standard Deviation); unit: events per hour] — The obstructive apnea-hypopnea index is similar to the standard AHI measure, but it only includes apnea or hypopnea events that are attributable to airway obstruction, as opposed to an origin in the central nervous system (referred to as "central sleep apnea"). This value reflects the numbers of times per hour the subject experienced an obstruction-related apnea or hypopnea event during sleep.
  events per hour | 22.0 (9.8)
Baseline central apnea index [Mean (Standard Deviation); unit: events per hour] — The central apnea-hypopnea index is similar to the standard AHI measure, but it only includes apnea or hypopnea events that arise from the central nervous system. Central apnea and hypopnea events are not caused by airway obstruction. This value reflects the numbers of times per hour the subject experienced a neurologically-related apnea or hypopnea event during sleep.
  events per hour | 1.6 (1.7)
Baseline hypopnea percentage [Mean (Standard Deviation); unit: percent (%)] — The hypopnea percentage describes the relative frequency of hypopnea events versus apnea events. Hypopnea is defined as shallow breathing, while apnea is defined as short pauses in breathing. The hypopnea percentage reflects what percentage of the total AHI can be attributed to hypopneas as opposed to apneas during sleep.
  percent (%) | 74.5 (32.2)
Baseline oxygenation percentage of SpO2 < 90% [Mean (Standard Deviation); unit: percent (%)] — During the overnight sleep studies, subjects' blood oxygen saturation (SpO2) were continuously monitored. This value reflects the percentage of their entire sleep time that the participants' blood oxygen saturation was below 90%.
  percent (%) | 1.4 (2.8)
Baseline SpO2 Nadir [Mean (Standard Deviation); unit: percent (%)] — The SpO2 nadir is the lowest blood oxygen saturation measurement taken throughout the sleep study.
  percent (%) | 84.6 (5.7)
Baseline percentage of time ETCO2 > 50 mmHg [Mean (Standard Deviation); unit: percent (%)] — End Tidal CO2 (ETCO2) is a measure of the carbon dioxide that is released at the end of a breath. Higher-than-normal end tidal CO2 measurements may be indicative of hypoventilation. We report here the percentage of time during sleep that subjects' end tidal CO2 exceeded the typical range of 50 mmHg.
  percent (%) | 21.8 (26.1)
Baseline sleep efficiency [Mean (Standard Deviation); unit: percent (%)] | 74.8 (16.8)
Baseline REM percentage [Mean (Standard Deviation); unit: percent (%)] | 12.8 (7.5)
Baseline arousal index [Mean (Standard Deviation); unit: events per hour] | 22.4 (11.1)
Baseline body mass index (BMI) [Count of Participants; unit: Participants]
  Normal (<85th percentile) | 23
  Overweight (85th to 95th percentile) | 19

OUTCOME MEASURES:

1. Primary Outcome: Serious Adverse Events
Description: In this study, adverse events were defined as "serious" if they resulted in: (1) death; (2) a life-threatening experience; (3) in-patient hospitalization or prolongation of hospital stay; (4) a persistent or significant disability/incapacity; (5) congenital anomaly/birth defect; or (6) events that jeopardized the health of the subject or required surgical intervention.
Time Frame: 1 year
Measure: Number; unit: participants
Groups:
- Inspire® Upper Airway Simulation System: Following hypoglossal nerve stimulator implantation, participants returned for a 1-week postoperative follow-up visit with their pediatric otolaryngologist. Titration polysomnography was performed 1, 3, 6, and 12 months after implantation. Quality-of-life assessments were completed at baseline and 12 months postoperatively. Adverse events were queried at every scheduled postoperative visit.
Arm/Group | Inspire® Upper Airway Simulation System
Number analyzed (Participants) | 42
participants | 7

2. Primary Outcome: Non-Serious Adverse Events
Description: Non-serious adverse events include all other adverse events recorded during the study which were determined to be related or possibly related to the device, surgery, or research. It does not include adverse events that were determined to be serious, as previously defined. Safety events that were determined to be unrelated to the study were not included in this analysis.
Time Frame: 1 year
Measure: Number; unit: participants
Arm/Group | Inspire® Upper Airway Simulation System
Number analyzed (Participants) | 42
participants | 15

3. Primary Outcome: Unanticipated Adverse Device Effects (UADE)
Description: Unanticipated adverse device effects (UADEs) are defined as adverse events which were determined to be serious, unexpected and related or possibly related to the investigational device.
Time Frame: 1 year
Measure: Number; unit: participants
Groups:
- Inspire® Upper Airway Simulation System: Following hypoglossal nerve stimulator implantation, participants returned for follow-up study visits 1 week, 1 month, 2 months, 6 months, and 12 months postoperatively. Adverse events were queried from the time of enrollment to the time of completing the 12 month visit.
Arm/Group | Inspire® Upper Airway Simulation System
Number analyzed (Participants) | 42
participants | 0

4. Secondary Outcome: Apnea-hypopnea Index (AHI)
Description: The apnea-hypopnea index (AHI) is a measure of the number of times per hour that an apnea or hypopnea event occurs during sleep. Apneas are defined as short pauses in breathing, while hypopnea is defined as shallow breathing. The AHI is useful in evaluating obstructive sleep apnea (OSA). The normal pediatric range is typically defined as an AHI of less than 1 event per hour. An AHI between 5 and 10 events per hour is consistent with moderate OSA, while an AHI above 10 suggests severe OSA. We report the mean AHI measured 1 year after device implantation. We also report the mean change in AHI, which compares AHI from baseline to 1 year postoperatively; therefore, negative change scores indicate a decrease from baseline to 1 year.
Time Frame: 1 year
Population: The analysis population includes all 42 participants who underwent hypoglossal nerve stimulator implantation. The 12 Month AHI was measured approximately 12 months following device implantation.
Measure: Mean (Standard Deviation); unit: events per hour
Groups:
- Inspire® Upper Airway Simulation System: Following hypoglossal nerve stimulator implantation, participants returned for a 1-week postoperative follow-up visit with their pediatric otolaryngologist. Titration polysomnography was performed 1, 3, 6, and 12 months after implantation. Quality-of-life assessments were completed at baseline and 12 months postoperatively.
Arm/Group | Inspire® Upper Airway Simulation System
Number analyzed (Participants) | 42
events per hour
  12 Month AHI | 11.0 (13.4)
  Change in AHI | -12.9 (13.2)
Statistical Analysis 1: Comparison: Inspire® Upper Airway Simulation System; Test type: Superiority; p < 0.0001, t-test, 2 sided

5. Secondary Outcome: Obstructive Apnea-hypopnea Index
Description: The obstructive apnea-hypopnea index is similar to the standard AHI measure, but it only includes apnea or hypopnea events that are attributable to airway obstruction, as opposed to an origin in the central nervous system (referred to as "central sleep apnea"). This value reflects the numbers of times per hour the subject experienced an obstruction-related apnea or hypopnea event during sleep. We report the mean obstructive AHI measured 1 year after device implantation. We also report the mean change in obstructive AHI, which compares obstructive AHI from baseline to 1 year postoperatively; therefore, negative change scores indicate a decrease from baseline to 1 year.
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: events per hour
Groups:
- Inspire® Upper Airway Simulation System: Following hypoglossal nerve stimulator implantation, titration polysomnography was performed 1, 2, 6, and 12 months after implantation.
Arm/Group | Inspire® Upper Airway Simulation System
Number analyzed (Participants) | 42
events per hour
  12 month obstructive apnea-hypopnea index | 10.1 (12.9)
  Change in obstructive apnea-hypopnea index | -12.2 (12.7)
Statistical Analysis 1: Comparison: Inspire® Upper Airway Simulation System; Test type: Superiority; p < 0.0001, t-test, 2 sided

6. Secondary Outcome: Central Apnea Index
Description: The central apnea-hypopnea index is similar to the standard AHI measure, but it only includes apnea or hypopnea events that arise from the central nervous system. Central apnea and hypopnea events are not caused by airway obstruction. This value reflects the numbers of times per hour the subject experienced a neurologically-related apnea or hypopnea event during sleep. We report the mean central apnea index measured 1 year after device implantation. We also report the mean change in central apnea index, which compares central apnea index from baseline to 1 year postoperatively; therefore, negative change scores indicate a decrease from baseline to 1 year.
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: events per hour
Arm/Group | Inspire® Upper Airway Simulation System
Number analyzed (Participants) | 42
events per hour
  12 month central apnea index | 0.87 (1.2)
  Change in central apnea index | -0.71 (1.7)
Statistical Analysis 1: Comparison: Inspire® Upper Airway Simulation System; Test type: Superiority; p = 0.035, t-test, 2 sided

7. Secondary Outcome: Hypopnea Percentage
Description: The hypopnea percentage describes the relative frequency of hypopnea events versus apnea events. Hypopnea is defined as shallow breathing, while apnea is defined as short pauses in breathing. The hypopnea percentage reflects what percentage of the total AHI can be attributed to hypopneas as opposed to apneas during sleep. We report the mean hypopnea percentage measured 1 year after device implantation. We also report the mean change in hypopnea percentage, which compares hypopnea percentage from baseline to 1 year postoperatively; therefore, negative change scores indicate a decrease from baseline to 1 year.
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: percent (%)
Arm/Group | Inspire® Upper Airway Simulation System
Number analyzed (Participants) | 42
percent (%)
  12 month hypopnea proportioin | 80.3 (21.9)
  Change in hypopnea proportion | 5.6 (33.9)
Statistical Analysis 1: Comparison: Inspire® Upper Airway Simulation System; Test type: Superiority; p = 0.083, t-test, 2 sided

8. Secondary Outcome: Oxygenation Percentage of Time SpO2 < 90%
Description: During the overnight sleep studies, subjects' blood oxygen saturation (SpO2) were continuously monitored. This value reflects the percentage of their entire sleep time that the participants' blood oxygen saturation was below 90%. We report the mean percentage of time SpO2 < 90% measured 1 year after device implantation. We also report the mean change in this time, which compares percentage of time from baseline to 1 year postoperatively; therefore, negative change scores indicate a decrease from baseline to 1 year.
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: percent (%)
Arm/Group | Inspire® Upper Airway Simulation System
Number analyzed (Participants) | 42
percent (%)
  12 month oxygenation percentage of time SpO2 < 90% | 0.6 (1.8)
  Change in oxygenation percentage of time SpO2 < 90% | -0.8 (3.1)
Statistical Analysis 1: Comparison: Inspire® Upper Airway Simulation System; Test type: Superiority; p = 0.0021, t-test, 2 sided

9. Secondary Outcome: Percentage of Time ETCO2 > 50 mmHg
Description: End Tidal CO2 (ETCO2) is a measure of the carbon dioxide that is released at the end of a breath. Higher-than-normal end tidal CO2 measurements may be indicative of hypoventilation. We report here the percentage of time during sleep that subjects' end tidal CO2 exceeded the typical range of 50 mmHg. We report the mean percentage of time measured 1 year after device implantation. We also report the mean change in percentage of time ETCO2 > 50 mmHg, which compares percentage of time from baseline to 1 year postoperatively; therefore, negative change scores indicate a decrease from baseline to 1 year.
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: percent (%)
Arm/Group | Inspire® Upper Airway Simulation System
Number analyzed (Participants) | 42
percent (%)
  12 month percentage of time ETCO2 > 50 mmHg | 14.0 (23.3)
  Change in percentage of time ETCO2 > 50 mmHg | -3.0 (31.5)
Statistical Analysis 1: Comparison: Inspire® Upper Airway Simulation System; Test type: Superiority; p = 0.764, t-test, 2 sided

10. Secondary Outcome: SpO2 Nadir
Description: The SpO2 nadir is the lowest blood oxygen saturation measurement taken throughout the sleep study. Change in SpO2 Nadir is defined from baseline to 1 year postoperatively; therefore, negative change scores indicate a decrease over time.
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: percent (%)
Arm/Group | Inspire® Upper Airway Simulation System
Number analyzed (Participants) | 42
percent (%)
  12 month SpO2 Nadir | 88.0 (4.5)
  Change in SpO2 Nadir | 3.2 (4.6)
Statistical Analysis 1: Comparison: Inspire® Upper Airway Simulation System; Test type: Superiority; p < 0.0001, t-test, 2 sided

11. Secondary Outcome: Sleep Efficiency
Description: Sleep efficiency is a measure of how much time that is dedicated to sleep is actually spent sleeping. Sleep efficiency is proportional to the amount of time spent asleep divided by the amount of time dedicated to sleep. Change in sleep efficiency is defined from baseline to 1 year postoperatively; therefore, negative change scores indicate a decrease over time.
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: percent (%)
Arm/Group | Inspire® Upper Airway Simulation System
Number analyzed (Participants) | 42
percent (%)
  12 month sleep efficiency | 72.2 (18.7)
  Change in sleep efficiency | -2.3 (19.7)
Statistical Analysis 1: Comparison: Inspire® Upper Airway Simulation System; Test type: Superiority; p = 0.467, t-test, 2 sided

12. Secondary Outcome: REM Percentage
Description: REM percentage is the percentage of sleep time that the participant spent in the rapid eye movement (REM) phase of sleep. Change in REM percentage is defined from baseline to 1 year postoperatively; therefore, negative change scores indicate a decrease over time.
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: percent (%)
Arm/Group | Inspire® Upper Airway Simulation System
Number analyzed (Participants) | 42
percent (%)
  12 month REM percentage | 13.2 (7.3)
  Change in REM percentage | 0.4 (8.8)
Statistical Analysis 1: Comparison: Inspire® Upper Airway Simulation System; Test type: Superiority; p = 0.745, t-test, 2 sided

13. Secondary Outcome: Arousal Index
Description: The arousal index measures the number of times per hour that the participant awoke from sleep. Change in arousal index is defined from baseline to 1 year postoperatively; therefore, negative change scores indicate a decrease over time.
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: events per hour
Arm/Group | Inspire® Upper Airway Simulation System
Number analyzed (Participants) | 42
events per hour
  12 month arousal index | 22.6 (20.1)
  Change in arousal index | -2.0 (19.7)
Statistical Analysis 1: Comparison: Inspire® Upper Airway Simulation System; Test type: Superiority; p = 0.106, t-test, 2 sided

14. Secondary Outcome: OSA-18 Total Survey Score
Description: The OSA-18 generates from participant responses a total score between 18 and 126 which is designed to reflect the impact of obstructive sleep apnea on the pediatric patient's quality of life. Higher total scores on the OSA-18 indicate a greater, negative impact on quality of life; while lower scores indicate a lesser impact on quality of life. Interpretation of total scores is as follows: minimal OSA impact for scores under 60; moderate OSA impact for scores between 60 and 80; and severe OSA impact for scores above 80. Change in OSA-18 total survey score is defined from baseline to 1 year postoperatively; therefore, negative change scores indicate a decrease of symptom severity over time.
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Inspire® Upper Airway Simulation System: The quality of life instruments (OSA-18 and Epworth Sleepiness Scale [ESS]) were administered at baseline (preoperatively) and 12 months postoperatively.
Arm/Group | Inspire® Upper Airway Simulation System
Number analyzed (Participants) | 42
units on a scale
  12 month OSA-18 total survey score | 31.3 (10.8)
  Change in OSA-18 total survey score | -34.8 (20.3)
Statistical Analysis 1: Comparison: Inspire® Upper Airway Simulation System; Test type: Superiority; p < 0.0001, t-test, 2 sided

15. Secondary Outcome: OSA-18 Overall Quality of Life Score
Description: The OSA-18 questionnaire includes a stand-alone question that asks to rate the child's overall quality of life on a scale from 0 (indicating worst quality of life possible) to 10 (indicating best quality of life possible). Change in OSA-18 overall score is defined from baseline to 1 year postoperatively; therefore, positive change scores indicate an improvement in quality of life over time.
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Inspire® Upper Airway Simulation System
Number analyzed (Participants) | 42
units on a scale
  12 month OSA-18 overall quality of life score | 8.1 (1.5)
  Change in OSA-18 overall quality of life score | 2.8 (1.9)
Statistical Analysis 1: Comparison: Inspire® Upper Airway Simulation System; Test type: Superiority; p < 0.0001, t-test, 2 sided

16. Secondary Outcome: Epworth Sleepiness Scale (ESS) Survey Score
Description: The ESS is a validated survey of daytime sleepiness. The ESS is scored as the sum of all items with scores ranging from 0 to 24 and higher scores indicating worse symptoms. Change ESS survey score is defined from baseline to 1 year postoperatively; therefore, negative change scores indicate an improvement in symptom severity over time.
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Inspire® Upper Airway Simulation System
Number analyzed (Participants) | 42
units on a scale
  12 month Epworth Sleepiness Scale (ESS) Survey Score | 5.0 (4.9)
  Change in Epworth Sleepiness Scale (ESS) Survey Score | -5.1 (6.9)
Statistical Analysis 1: Comparison: Inspire® Upper Airway Simulation System; Test type: Superiority; p < 0.0001, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Participants were monitored for adverse events for 1 year following hypoglossal nerve stimulator implantation.
Arm/Group | Inspire® Upper Airway Simulation System
All-Cause Mortality (participants affected / at risk) | 0/42
Serious Adverse Events (participants affected / at risk) | 7/42
Other Adverse Events (participants affected / at risk) | 15/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Inspire® Upper Airway Simulation System (N=42)
Hospitalization for postoperative pain or discomfort (General disorders) | 3 (3) — Three (3) participants were hospitalized for postoperative pain or discomfort. Duration of hospital stay for this reason ranged from 2 to 5 nights. The SAE resolved without sequelae in all 3 participants.
Prolonged surgical duration (Surgical and medical procedures) | 1 (1) — Due to anatomical complexity, one (1) participant's implantation surgery was prolonged, resulting in erythema and parietal tenderness for 1 week following surgery. This SAE resolved without sequelae.
Surgical revision (Surgical and medical procedures) | 2 (2) — Two (2) participants required surgical revisions to fix a lead connection issue and to correct a lead protrusion through the submental incision. Both SAEs resolved without sequelae.
Not related to device, surgery, or research (General disorders) | 2 (2) — Two (2) participants experienced serious adverse events during the course of the study that were deemed unrelated to the device, surgery, or research.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Inspire® Upper Airway Simulation System (N=42)
Tongue/oral pain or discomfort (Surgical and medical procedures) | 5 (6)
Rash at surgical site (Skin and subcutaneous tissue disorders) | 4 (4)
Acute insomnia (Nervous system disorders) | 2 (3)
Cellulitis at surgical site (Skin and subcutaneous tissue disorders) | 2 (2)
Cheek swelling (Skin and subcutaneous tissue disorders) | 1 (1)
Forehead abscess from PSG electrodes (Skin and subcutaneous tissue disorders) | 1 (1)
Perioperative urinary retention (Renal and urinary disorders) | 1 (1)
Post-obstructive central hypoventilation (Respiratory, thoracic and mediastinal disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Analysis was limited by the lack of a control group, although spontaneous resolution of OSA would be less likely to occur in an adolescent population with severe disease. Not all of the 12-month PSGs were full-night studies at one voltage. Some of the patients were young adults over 18 years old, and there are different scoring criteria for adolescents compared to young adults. All patients were assessed using the same criteria in order to maintain consistency across the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2020-05-08): https://cdn.clinicaltrials.gov/large-docs/08/NCT02344108/Prot_000.pdf
  • Informed Consent Form (2019-11-08): https://cdn.clinicaltrials.gov/large-docs/08/NCT02344108/ICF_001.pdf